CLINICAL TRIAL: NCT00406380
Title: Does Avastin Change Evolution in Juxtafoveal Telangiectasias?
Brief Title: Effect of Avastin in Juxtafoveal Telangiectasias
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: APEC-0024
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Telangiectasis
Keywords: Telangiectasias; Leakage; Bevacizumab; Telangiectasias secondary to Branch Retinal Vein Occlusion (BRVO); Idiopathic juxtafoveal retinal telangiectasias
MeSH Terms: conditions — Telangiectasis | interventions — Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab
Procedure: Intravitreal injection of Bevacizumab

SUMMARY:
Evaluation of efficacy of Intravitreal Injection of Bevacizumab in patients with Yuxtafoveal Telangiectasias

DETAILED DESCRIPTION:
After diagnose Yuxtafoveal telangiectasias secondary to Branch Retinal Vein Occlusion and with Idiopathic Ethiology by clinical signs and Fluorescein angiogram (FA)findings we treated patients with Intravitreal Injection of Bevacizumab (2.5mg/0.1ml). We performed a complete ophthalmological evaluation and at baseline and follow-up (1 and 3 months) we evaluate ETDRS Best Corrected visual acuity (BCVA), fluorescein angiogram (FA) and Optical Coherence Tomography (OCT)findings. We found an improvement in visual acuity and reduction of FA leakage and decrease retinal thickness in OCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Telangiectasias secondary to Branch Retinal Vein Occlusion
* Patients with Idiopathic Juxtafoveal Retinal Telangiectasias

Exclusion Criteria:

* Diabetic Retinopathy and Diabetic Macular Edema
* Hypertensive Retinopathy
* Choroidal Neovascularization

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2006-09 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Best corrected Visual Acuity
Fluorescein Angiogram: Leakage
Optical Coherence Tomography: Retinal thickness

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Kon-Jara, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociacion para Evitar la Ceguera en Mexico, Mexico City, Mexico City, Mexico